CLINICAL TRIAL: NCT07208149
Title: A Phase Ib/IIa, Open-Label, Two-Cohort, Dose-Escalation and Dose-Expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of MR001 in Patients With Locally Recurrent or Metastatic Advanced Triple-Negative Breast Cancer (TNBC) Who Have Progressed After First-Line or Later-Line Therapy
Brief Title: A Study of MR001 in Patients With Locally Recurrent or Metastatic Advanced Triple-Negative Breast Cancer (TNBC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Majory Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MJR-MR001-03
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Triple-Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose Escalation Part, Dose Group A: MR001 1 mg/kg, QW (Experimental)
  Interventions: Drug: MR001 Bispecific Antibody for Injection
- Dose Escalation Part, Dose Group B: MR001 2 mg/kg, QW (Experimental)
  Interventions: Drug: MR001 Bispecific Antibody for Injection
- Dose Escalation Part, Dose Group C: MR001 4 mg/kg, QW (Experimental)
  Interventions: Drug: MR001 Bispecific Antibody for Injection
- Dose Escalation Part, Dose Group D: MR001 2 mg/kg, Q2W (Experimental)
  Interventions: Drug: MR001 Bispecific Antibody for Injection
- Dose Expansion Part (Experimental): Based on the Dose escalation part results, the Investigator and Sponsor will determine one dose and dosing interval to proceed to the dose expansion study
  Interventions: Drug: MR001 Bispecific Antibody for Injection

INTERVENTIONS:
Drug: MR001 Bispecific Antibody for Injection — Intravenous infusion

SUMMARY:
This Phase Ib/IIa study is evaluating the safety, tolerability, pharmacokinetics, and preliminary efficacy of MR001 in patients with advanced triple-negative breast cancer (TNBC) who have progressed after prior therapy.

DETAILED DESCRIPTION:
This is a dual-cohort, open-label, dose escalation and dose expansion Phase Ib/IIa study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-tumor activity of MR001 in patients with locally recurrent or metastatic advanced triple-negative breast cancer (TNBC) who have progressed after first-line or later-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed triple-negative breast cancer (TNBC).
* Subjects with locally recurrent or metastatic advanced TNBC who have progressed after first-line or later-line therapy.
* Presence of at least one measurable lesion according to RECIST V1.1 criteria.
* ECOG Performance Status 0 or 1.
* Life expectancy >3 months.
* Adequate organ and hematopoietic function based on the laboratory tests.
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* History of severe allergy or hypersensitivity to the investigational product or its excipients or drugs of similar chemical class (e.g., monoclonal antibodies), or contraindications to the investigational product.
* Requirement for systemic immunosuppressive therapy within 14 days prior to the first dose of study drug or during the study.
* Major surgery (excluding puncture biopsy) within 4 weeks prior to the first dose of study drug, or anticipated need for major surgery during this study.
* Uncontrolled active brain metastases or leptomeningeal metastasis.
* History of autoimmune disease requiring treatment with corticosteroids or immunosuppressive drugs.
* Women in the period of preconception, pregnancy, or lactation.
* Any other circumstances which the investigator considers may increase risks to subjects or interfere with the results of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience one or more dose-limiting toxicities (DLTs) | Approximately 6 months
Maximum Tolerated Dose (MTD) of MR001 | Approximately 6 months
  The maximum tolerated dose (MTD) of MR001 was assessed for QW dosing schedules
Incidence of Adverse Events (AEs) as Assessed by CTCAE v5.0 | Approximately 2 years

SECONDARY OUTCOMES:
Recommended Phase II Dose (RP2D) based on safety, pharmacodynamics, pharmacokinetics and Preliminary Anti-tumor Activity of MR001 | Approximately 6 months
Progression-free survival (PFS) | Approximately 2 years
Duration of response (DOR) | Approximately 2 years
Overall survival (OS) | Approximately 3 years
Objective Response Rate (ORR) | Approximately 2 years
Area Under the Plasma Concentration-Time Curve (AUC) of MR001 | Predose and at designated timepoints in each cycle for approximately 2 years (each cycle = 2 weeks)
Maximum Plasma Concentration (Cmax) of MR001 | Predose and at designated timepoints in each cycle for approximately 2 years (each cycle = 2 weeks)
Time to Maximum Plasma Concentration (Tmax) of MR001 | Predose and at designated timepoints in each cycle for approximately 2 years (each cycle = 2 weeks)
Change from baseline at different time points for TGF-β1 in plasma | Predose and at designated timepoints during the first three cycles (each cycle = 2 weeks)
Change from baseline at different timepoints for Th1 of MR001 | Predose and at designated timepoints during the first three cycles (each cycle = 2 weeks)
Change from baseline at different timepoints for Th2 of MR001 | Predose and at designated timepoints during the first three cycles (each cycle = 2 weeks)
Incidence of Antidrug Antibodies (ADA) to MR001 | Predose in each cycle for approximately 2 years (each cycle = 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China